CLINICAL TRIAL: NCT01968278
Title: Use of Baked Milk in Oral Immunotherapy for Severe IgE-mediated Cow's Milk Protein Allergic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Assaf Harofeh MC, Helsinki commitee, Assaf-Harofeh Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 39/12 Asaf
Record Dates: First submitted 2013-08-25; First posted 2013-10-24 (Estimated); Last update posted 2013-10-24 (Estimated); Status verified 2013-10

CONDITIONS: Cow's Milk Allergy
MeSH Terms: conditions — Milk Hypersensitivity

ARMS (2):
- Baked milk group (Experimental): BM (baked milk)
  Interventions: Other: Baked milk
- Control (No Intervention): IgE-cow's milk allergic patients not treated with OIT

INTERVENTIONS:
Other: Baked milk
  Arms: Baked milk group

SUMMARY:
Oral immunotherapy (OIT) programs for milk, egg and peanut, desensitize patients to their respective allergens and thereby decrease their risk of morbidity and mortality. OIT programs, however, are not without adverse events, particularly in highly sensitive patients. Recently, it has been demonstrated that the administration of baked milk (BM) products to IgE-CMA patients that are non-reactive to BM, can promote tolerance to unheated milk (UM). The goal of our research is to determine whether BM can promote desensitization even in the highly sensitive patient, who reacts to baked milk as well. In a second step, we hypothesize BM-OIT will promote desensitization to unheated milk, as well.

Importance: The change in the risk/benefit ratio of such a program will alter the therapeutic approach to an IgE-CMP allergic patient.

Probable implications to Medicine: BM-OIT will allow highly sensitive patients to tolerate milk products, decreasing their risk of life-threatening reactions. Furthermore, analysis of the immune modulation parameters that change during the treatment program, should pave the way for defining mechanisms underlying tolerance in CMP allergy.

DETAILED DESCRIPTION:
In our first aim, we will test over a four day induction (escalating) program, whether highly sensitive UM-reactive patients) can tolerate BM . Those successful will be randomized to a treated BM-OIT group (group A) and an observational control group (group B). In the second aim, the fraction of patients in Group A who successfully progress in BM-OIT (tolerate ≥ 360 mg BM) over a 6 month period will be determined and compared to the fraction of patients in Group B who can tolerate 360mg. The results will also be compared to the progression of highly sensitive IgE-CMA patients on UM-OIT (Group C, reactive to ≤21 mg of UM ). In aim-3, the fraction of BM-OIT patients able to tolerate minimally ≥ 12.5 mg of UM or higher than their initially eliciting dose. will be assessed.

Methods: Severe patients (>4 years) with a positive clinical history, SPT and a positive DBPCFC to CMP will be first tested for their ability to tolerate BM. The treatment group will undergo three rounds of oral induction, each consisting of 4 days and performed every 4 weeks. On day #1, the patient will be rapidly desensitized up to their threshold. On days 2-3, the maximum tolerable dose and interval is determined. Day #4 mimics the home treatment. Home treatment will then continue until the next induction. After 6 months of treatment patients will be evaluated for reactivity to UM.

ELIGIBILITY:
Inclusion Criteria:

Patients with IgE-cow's milk allergy reacting to <12.5 mg (any reaction) on oral food challenge to unheated milk

Exclusion Criteria:

Patients with unstable asthma** or those with suspected compliance issues will be excluded. Patients with stable asthma are included.

* defined as active wheezing and/or use of oral steroids within one month prior to initiation of program and/or FEV1<75% or a greater than 18% increase in FEV1 after bronchodilator treatment.

Ages: 4 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
The amount of milk protein (mg) that can be tolerated as baked milk in highly sensitized CMA patietns | Day 1

SECONDARY OUTCOMES:
The increase in tolerated CMP (mg) following 6 month of OIT in comparison to an observational control group kept on a CMP free diet | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Asaf Harofeh Medical Center, Beer Yaakoc, Zerifin, Israel

REFERENCES:
- [Derived] Goldberg MR, Nachshon L, Appel MY, Elizur A, Levy MB, Eisenberg E, Sampson HA, Katz Y. Efficacy of baked milk oral immunotherapy in baked milk-reactive allergic patients. J Allergy Clin Immunol. 2015 Dec;136(6):1601-1606. doi: 10.1016/j.jaci.2015.05.040. Epub 2015 Jul 17. PMID 26194541